CLINICAL TRIAL: NCT00565643
Title: A Multicenter, Randomized, Controlled Trial of Seprafilm® Adhesion Barrier to Reduce Adhesion Formation Following Cesarean Delivery
Brief Title: Seprafilm® Adhesion Barrier and Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Collaborators: Stony Brook University (Other); Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Daniel Kiefer, Principal Investigator, Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB No. 07023; MO1RR10710 (Other Grant/Funding Number: General Clinical Research Center (GCRC))
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Adhesions; Cesarean Section; Delivery, Obstetric
Keywords: Adhesion; Seprafilm; Cesarean section
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HA-CMC Group (Experimental): Hyaluronic Acid-Carboxymethylcellulose placed as an adhesion barrier
  Interventions: Device: modified sodium hyaluronic acid and carboxymethylcellulose
- Routine Closure Group (Placebo Comparator): Routine Closure without placement of an adhesion barrier
  Interventions: Device: Placebo

INTERVENTIONS:
Device: modified sodium hyaluronic acid and carboxymethylcellulose — Adhesion barrier applied at the time of initial cesarean delivery
  Other Names: Seprafilm Adhesion Barrier
  Arms: HA-CMC Group
Device: Placebo — Routine abdominal closure without placement of adhesion barrier
  Arms: Routine Closure Group

SUMMARY:
A multicenter, randomized, controlled, single blinded study to evaluate the effectiveness of Seprafilm® Adhesion Barrier in reducing adhesion formation in cesarean deliveries. Primary outcome will be measurement of the extent and severity of adhesions at the time of subsequent cesarean delivery. Secondary outcomes will include measures of safety, operative times (ex., incision-delivery; total operative time).

DETAILED DESCRIPTION:
Patients presenting to labor and delivery for delivery will be screened for eligibility. If a patient meets the inclusion and exclusion criteria, she will be offered enrollment in the study. After the project and informed consent are reviewed with the patient and all questions are answered, she will be asked to sign the informed consent. At this point, she will be considered a candidate for randomization.

If the patient subsequently undergoes a cesarean delivery, she will be randomized to either:

1. Group A - Placement of Seprafilm® prior to abdominal closure
2. Group B - Routine closure without placement of Seprafilm® The chances of being assigned to either group will be equal (i.e., 1:1 randomization). The patient will be blinded with regard to Seprafilm placement.

The investigators will collect additional data about the patient, her antepartum course, intra-operative events, and post-operative course. There are no additional tests or procedures ordered or performed during the hospital stay as part of this protocol. Enrollment in this study is not expected to alter the patient's length of stay.

The antepartum, operative, and post-operative care of the patient will as directed by the patient's physician and participating institutions's standard policies and procedures. This study in no way changes or directs the care the patient would receive, except with regard to the placement of Seprafilm® Adhesion Barrier.

A short-term telephone follow-up will be conducted approximately 6-8 weeks following randomization to assess for immediate post-operative complications.

If a patient becomes pregnant again and undergoes a repeat cesarean delivery at a participating institution, the location and severity of adhesions (if any) would be assessed at the time of repeat cesarean delivery. The investigators will extract additional data from the chart including operative times, blood loss, and complications. An evaluation of adhesions would conclude the patient's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are planning or have the potential to undergo cesarean delivery
* Age over 18
* Able to consent to study

Exclusion Criteria:

* Planned tubal ligation
* Known allergy to hyaluronic acid
* Medical or other serious condition which will interfere with compliance and/or ability to complete study protocol

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 753 (Actual)
Dates: Start 2007-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Kiefer, M.D., Principal Investigator — Lehigh Valley Health Network
Locations (3):
- United States (3):
  - Winthrop University Hospital, Mineola, New York
  - SUNY Stony Brook University Hospital, Stony Brook, New York
  - Lehigh Valley Hospital, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HA-CMC Group: modified sodium hyaluronic acid and carboxymethylcellulose (Seprafilm Adhesion Barrier): Adhesion barrier applied at the time of cesarean delivery
Period: Overall Study
Arm/Group | HA-CMC Group | Routine Closure Group
Started | 380 | 373
Safety Data | 380 | 373
Primary Outcome (Subsequent Cesarean) | 80 | 92
Completed | 380 | 373
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HA-CMC Group | Routine Closure Group | Total
Number analyzed (Participants) | 380 | 373 | 753
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.1) | 30.9 (5.3) | NA (NA) — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 380 | 373 | 753
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 380 | 373 | 753
Gravid [Mean (Full Range); unit: pregnancies] | 2 [1 to 20] | 2 [1 to 11] | NA [NA to NA] — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
Parity [Median (Full Range); unit: pregnancies] | 1 [0 to 4] | 1 [0 to 4] | NA [NA to NA] — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
Gestational age (weeks) [Mean (Standard Deviation); unit: weeks] | 38.7 (1.9) | 38.1 (3.9) | NA (NA) — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
Body Mass Index (BMI), kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 33.3 (6.6) | 33.2 (7.8) | NA (NA) — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
# of previous cesarean births [Median (Full Range); unit: births] | 1 [0 to 3] | 1 [0 to 3] | NA [NA to NA] — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
Preoperative Hematocrit [Mean (Standard Deviation); unit: percent] | 34.8 (4.3) | 34.4 (5.0) | NA (NA) — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
Preoperative White Blood cell count [Mean (Standard Deviation); unit: cells/mm^3] | 10.3 (3.4) | 10.7 (4.6) | NA (NA) — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.
Preoperative Maximum Temperature [Mean (Standard Deviation); unit: degrees Fahrenheit] | 97.8 (1.0) | 97.9 (0.9) | NA (NA) — The Totals are unable to be calculated because the analysis was not performed for the Total population and there are no means to calculate.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adhesions
Description: The Percentage of participants with one or more adhesions, regardless of the extent or severity
Time Frame: 3 to 5 years
Measure: Number; unit: percentage of patients with adhesions
Arm/Group | HA-CMC Group | Routine Closure Group
Number analyzed (Participants) | 80 | 92
percentage of patients with adhesions | 75.6 | 75.9

2. Secondary Outcome: Post-operative Hemoglobin
Description: Hemoglobin level following randomization delivery - used to determine if there was a difference in blood loss between the two groups
Time Frame: 1 to 5 years
Measure: Mean (Standard Deviation); unit: % of blood that is red blood cells
Arm/Group | HA-CMC Group | Routine Closure Group
Number analyzed (Participants) | 380 | 373
% of blood that is red blood cells | 29.9 (4.1) | 30.2 (3.6)

3. Primary Outcome: Adhesion Score
Description: Adhesion score. Derived by assigning 1 point for filmy adhesion and 2 points for dense adhesions at each of 6 possible sites in the abdomen. Thus the score can range from 0 (i.e., no adhesions at any location) to 12 (dense adhesions at each site).
Time Frame: 3 to 5 years
Measure: Median (Full Range); unit: units on a scale
Groups:
- HA-CMC Group: modified sodium hyaluronic acid and carboxymethylcellulose (Seprafilm Adhesion Barrier): Adhesion barrier applied at the time of initial cesarean delivery
Arm/Group | HA-CMC Group | Routine Closure Group
Number analyzed (Participants) | 80 | 92
units on a scale | 2 [0 to 10] | 2 [0 to 8]

4. Secondary Outcome: Post-operative White Blood Cell Count
Description: Post-operative White blood cell count following randomization delivery - used to determine if there was difference in immune response or infection between the groups
Time Frame: 1 to 5 years
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | HA-CMC Group | Routine Closure Group
Number analyzed (Participants) | 380 | 373
cells/mm^3 | 11.3 (6.4) | 11.0 (3.3)

5. Secondary Outcome: Post-Operative Complications
Description: Percentage of patients experiencing any of the predefined post-operative complications following randomization
Time Frame: 1 to 5 years
Measure: Number; unit: % of patients experiencing complication
Arm/Group | HA-CMC Group | Routine Closure Group
Number analyzed (Participants) | 380 | 373
% of patients experiencing complication
  Any complication | 6.3 | 4.0
  Fever | 4.5 | 3.0
  Ileus or bowel obstruction | 0 | 0
  Any wound complication | 2.1 | 0.8
  Venous thromboembolism | 0 | 0.3
  Readmission (<=6 weeks postpartum) | 1.3 | 0.5

6. Secondary Outcome: Post-operative Maximum Temperature Following Randomization
Description: Maximum temperature of patient, >24 hours following randomization delivery
Time Frame: 1 to 5 years
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | HA-CMC Group | Routine Closure Group
Number analyzed (Participants) | 380 | 373
degrees Fahrenheit | 98.2 (1.0) | 98.2 (0.9)

7. Secondary Outcome: Operative Times at Subsequent Delivery
Description: Amount of time spent at the time of the subsequent delivery
Time Frame: 3 to 5 years
Measure: Median (Full Range); unit: minutes
Arm/Group | HA-CMC Group | Routine Closure Group
Number analyzed (Participants) | 80 | 92
minutes
  Skin-to-delivery | 13 [3 to 70] | 13 [4 to 55]
  Total operative time | 51 [23 to 175] | 54 [26 to 157]

ADVERSE EVENTS:
Time Frame: From time of enrollment through 8 weeks following randomization
Arm/Group | HA-CMC Group | Routine Closure Group
Serious Adverse Events (participants affected / at risk) | 5/380 | 2/373
Other Adverse Events (participants affected / at risk) | 0/380 | 0/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HA-CMC Group (N=380) | Routine Closure Group (N=373)
Readmission for Infection (Infections and infestations) | 2 (2) | 1 (1)
Readmission for Intra-abdominal complication (Gastrointestinal disorders) | 2 (2) | 0 (0)
Readmission for Central nervous system problem (Nervous system disorders) | 0 (0) | 1 (1)
Readmission for obstetrical complications (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Delayed Postpartum hemorrhage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No